CLINICAL TRIAL: NCT01421017
Title: Phase I/II Study of TLR7 Agonist Imiquimod, Cyclophosphamide, and Radiotherapy in Breast Cancer Patients With Chest Wall Recurrence or Skin Metastases
Brief Title: Toll-like Receptor (TLR) 7 Agonist, Cyclophosphamide, and Radiotherapy for Breast Cancer With Skin Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-00598; 1R01CA161891-01 (NIH)
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: radiation therapy; combination therapy; immunotherapy; immune response modifier; immunostimulatory; immunomodulator
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation; Imiquimod; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- IMQ+RT (Experimental): This arm has been closed as of 6/4/2014.
  * Weeks 1-2: RT given to one metastatic skin site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W)
  * Weeks 1-8: day 1-5 of each week: imiquimod 5% cream applied to all skin sites overnight, starting on day 1 after RT, day 6-7 of each week: rest period.
  * Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Interventions: Radiation: Radiation; Drug: Imiquimod
- CTX/IMQ/RT (Experimental): * Week -1 (day-7): cyclophosphamide 200mg/m2 IV as single infusion
  * Weeks 1-2: RT given to one metastatic skin site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W)
  * Weeks 1-8: day 1-5 of each week: imiquimod 5% cream applied all sites overnight, starting on day 1 after RT, day 6-7 of each week: rest period.
  * Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Interventions: Radiation: Radiation; Drug: Imiquimod; Drug: Cyclophosphamide
- CTX/RT (Experimental): For patients with only non-skin metastatic sites
  First cycle (Cycle 1):
  * Week -1 (day -7): cyclophosphamide 200mg/m2 IV as single infusion
  * Weeks 1-2: RT given to one site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W)
  * Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Interventions: Radiation: Radiation; Drug: Cyclophosphamide

INTERVENTIONS:
Radiation: Radiation
Drug: Imiquimod
  Other Names: ALDARA
  Arms: CTX/IMQ/RT; IMQ+RT
Drug: Cyclophosphamide
  Other Names: Cytoxan
  Arms: CTX/IMQ/RT; CTX/RT

SUMMARY:
This study is to find an optimal dose of Imiquimod (IMQ) in the first part (Phase I) and test the effectiveness of the combination treatment of IMQ, cyclophosphamide (CTX), and radiotherapy (RT) in patients with skin metastases from breast cancer in the second part (Phase II). Currently this trial is in its Phase II part.

DETAILED DESCRIPTION:
By harnessing the cytocidal and immunostimulatory properties of two local treatment modalities, RT and IMQ, an effective, adaptive immune response can be generated, resulting in systemic control of metastatic breast cancer after local treatment of cutaneous metastases. Additionally, based on investigators' recent preclinical data, the investigators intend to estimate in patients with metastatic breast cancer, if the addition of immunomodulatory cyclophosphamide can increase anti-tumor responses.

This trial originally had one treatment arm IMQ/RT(patients were treated with IMQ and RT). Recent evidence has emerged that the addition of immunomodulatory cyclophosphamide (CTX) increased anti-tumor responses, therefore the IMQ/RT arm is closed and the trial will continue with two additional cohorts (CTX/IMQ/RT and CTX/RT) which include cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-confirmed breast cancer.
2. Patients with at least measurable skin metastases and distant, measurable metastases (outside of skin) by Response Evaluation Criteria in Solid Tumors (RECIST). For patients without distant measurable metastases, an area of the skin metastases designated to not receive local therapy can be substituted. Patients with multiple (>= 2) metastatic sites (skin involvement not required), with at least one site measurable by RECIST, will be eligible for the CTX/RT cohort.
3. Age >= 18 years.
4. Eastern Cooperative Oncology Group performance status 0-2.
5. Patients must agree to tumor fine-needle aspiration required by protocol.
6. Concurrent systemic cancer therapy (hormones, biologics or chemotherapy) can be continued if distant metastases are non-responsive (i.e. no complete response or partial response) on that regimen for >= 8 weeks as assessed by the investigator.
7. Patients must have adequate organ and bone marrow function as defined below:

   * absolute neutrophil count >= 1,300/microliter
   * hemoglobin >= 9.0 grams/deciliter
   * platelets >= 75,000/microliter
   * total bilirubin =< 1.5 X institutional upper limit of normal
   * AST (aspartate aminotransferase) =< 2.5 X institutional upper limit of normal
   * ALT (alanine aminotransferase) =< 2.5 X institutional upper limit of normal
   * creatinine =< 2 X institutional upper limit of normal if patient has chronic renal insufficiency and creatinine has been stable for > 4 months)
8. Informed consent.

Exclusion Criteria:

1. Brain metastases unless resected or irradiated and stable >= 4 weeks.
2. Concurrent treatment with other investigational agents.
3. Patients who have received any local therapy (radiotherapy, high-potency corticosteroids, intralesional therapy, laser therapy or surgery) other than biopsy to the target area within 4 weeks prior to first dosing of study agent.
4. Patients who have received hyperthermia to the target area within 10 weeks prior to first dosing of study agent.
5. Patients with an uncontrolled bleeding disorder.
6. Patients (with skin metastases only) who will be therapeutically anticoagulated with heparins or coumadin at the time of the biopsy (they are eligible if anticoagulation can be held prior to biopsy as per investigator). Patients on aspirin and other platelet agents are eligible.
7. Patients with known immunodeficiency or receiving immunosuppressive therapies.
8. History of allergic reactions to imiquimod or its excipients.
9. Uncontrolled intercurrent medical illness or psychiatric illness/social situations that would limit compliance with study requirements.
10. Pregnancy or lactation.
11. Women of childbearing potential not using a medically acceptable means of contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-08-19 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Adams, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Kouloulias VE, Dardoufas CE, Kouvaris JR, Gennatas CS, Polyzos AK, Gogas HJ, Sandilos PH, Uzunoglu NK, Malas EG, Vlahos LJ. Liposomal doxorubicin in conjunction with reirradiation and local hyperthermia treatment in recurrent breast cancer: a phase I/II trial. Clin Cancer Res. 2002 Feb;8(2):374-82. PMID 11839652
- [Derived] Adams S, Demaria S, Rinchai D, Wang E, Novik Y, Oratz R, Fenton-Kerimian M, Levine PG, Li X, Marincola F, Jin P, Stroncek D, Goldberg J, Bedognetti D, Formenti SC. Topical TLR7 agonist and radiotherapy in patients with metastatic breast cancer. J Immunother Cancer. 2025 Apr 5;13(4):e011173. doi: 10.1136/jitc-2024-011173. PMID 40187749

RESULTS

PARTICIPANT FLOW:
Groups:
- IMQ+RT: This arm has been closed as of 6/4/2014.
  * Weeks 1-2: RT given to one metastatic skin site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W)
  * Weeks 1-8: day 1-5 of each week: imiquimod 5% cream applied to all skin sites overnight, starting on day 1 after RT, day 6-7 of each week: rest period.
  * Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Radiation
  Imiquimod
- CTX/IMQ/RT: * Week -1 (day-7): cyclophosphamide 200mg/m2 IV as single infusion
  * Weeks 1-2: RT given to one metastatic skin site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W)
  * Weeks 1-8: day 1-5 of each week: imiquimod 5% cream applied all sites overnight, starting on day 1 after RT, day 6-7 of each week: rest period.
  * Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Radiation
  Imiquimod
  Cyclophosphamide
- CTX/RT: For patients with only non-skin metastatic sites
  First cycle (Cycle 1):
  * Week -1 (day -7): cyclophosphamide 200mg/m2 IV as single infusion
  * Weeks 1-2: RT given to one site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W)
  * Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Radiation
  Cyclophosphamide
Period: Overall Study
Arm/Group | IMQ+RT | CTX/IMQ/RT | CTX/RT
Started | 12 | 12 | 7
Completed | 10 | 6 | 4
Not Completed | 2 | 6 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — POD | 0 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMQ+RT | CTX/IMQ/RT | CTX/RT | Total
Number analyzed (Participants) | 12 | 12 | 7 | 31
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean Age | 67 (6.2) | 51 (7.4) | 51 (7.1) | 57 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 6 | 30
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 10 | 12 | 6 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 8 | 8 | 1 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Systemic Tumor Response Rates (Complete Response+Partial Response)
Description: The systemic tumor response refers to the response at the time of best overall response. The response criteria are specially adapted from Response Evaluation Criteria in Solid Tumor for Immunotherapies (Wolchok, et al., 2009).
Time Frame: 9 weeks from the start of the treatment of RT
Measure: Number (95% Confidence Interval); unit: proportion of tumors
Arm/Group | IMQ+RT | CTX/IMQ/RT | CTX/RT
Number analyzed (Participants) | 12 | 12 | 7
proportion of tumors | .25 [.06 to .57] | .083 [.002 to .38] | 0 [0 to 0]

2. Secondary Outcome: Local Skin Tumor Response Rates (Complete Response + Partial Response)
Description: The response refers to the best overall response, based on European Organization for Research and Treatment of Cancer's definitions for chest wall tumors (Kouloulias, et al., 2002).
Time Frame: 9 weeks from the start of the treatment
Population: Arm "CTX/RT" is not applicable, as it includes only patients with non-skin metastatic sites.
Measure: Number (95% Confidence Interval); unit: proportion of tumors
Arm/Group | IMQ+RT | CTX/IMQ/RT
Number analyzed (Participants) | 12 | 12
proportion of tumors
  Local Area A; irradiated area | 0.83 [.52 to .98] | 0.75 [.43 to .95]
  Local Area B; non-irradiated area | .33 [.10 to .65] | .083 [.002 to .38]

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- IMQ+RT: This arm has been closed as of 6/4/2014.
  Weeks 1-2: RT given to one metastatic skin site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W) Weeks 1-8: day 1-5 of each week: imiquimod 5% cream applied to all skin sites overnight, starting on day 1 after RT, day 6-7 of each week: rest period.
  Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Radiation Imiquimod
- CTX/IMQ/RT: Week -1 (day-7): cyclophosphamide 200mg/m2 IV as single infusion Weeks 1-2: RT given to one metastatic skin site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W) Weeks 1-8: day 1-5 of each week: imiquimod 5% cream applied all sites overnight, starting on day 1 after RT, day 6-7 of each week: rest period.
  Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Radiation Imiquimod Cyclophosphamide
- CTX/RT: For patients with only non-skin metastatic sites
  First cycle (Cycle 1):
  Week -1 (day -7): cyclophosphamide 200mg/m2 IV as single infusion Weeks 1-2: RT given to one site at 6 Gy on days 1, 3, 5, 8 and 10 (M-W-F-M-W) Week 9: response assessment
  Patients may continue to receive additional cycles (same schedule, RT given to a different site), provided that patients wish to continue, are without clinically significant progression and further treatment may be beneficial in the opinion of the investigator.
  Radiation Cyclophosphamide
Arm/Group | IMQ+RT | CTX/IMQ/RT | CTX/RT
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/12 | 1/7
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMQ+RT (N=12) | CTX/IMQ/RT (N=12) | CTX/RT (N=7)
Breast Infection (Infections and infestations) | 1 | 0 | 0
Breast Pain (General disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tumor Pain (General disorders) | 2 | 0 | 0
Neosplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Blurred Vision (Eye disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Headache (General disorders) | 0 | 1 | 0
Pain in extremity (General disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Adult respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMQ+RT (N=12) | CTX/IMQ/RT (N=12) | CTX/RT (N=7)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 12 | 0
Anemia (Blood and lymphatic system disorders) | 12 | 12 | 7
Anxiety (Psychiatric disorders) | 0 | 12 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 12 | 0
Back Pain (General disorders) | 0 | 12 | 0
Breast Pain (General disorders) | 12 | 12 | 0
Constipation (Gastrointestinal disorders) | 0 | 12 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 7
Depression (Psychiatric disorders) | 0 | 12 | 0
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 12 | 12 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 12 | 7
Dysarthria (Musculoskeletal and connective tissue disorders) | 0 | 12 | 0
Fatigue (General disorders) | 12 | 12 | 7
Headache (General disorders) | 0 | 12 | 0
Lymphedema (Blood and lymphatic system disorders) | 0 | 12 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 12 | 0
Nausea (General disorders) | 12 | 12 | 7
Pain (General disorders) | 12 | 12 | 0
Paresthesia (Musculoskeletal and connective tissue disorders) | 0 | 12 | 7
Abdominal Distension (Gastrointestinal disorders) | 12 | 0 | 7
Alkaline Phosphatase Increased (Gastrointestinal disorders) | 0 | 0 | 7
Aspartate Aminotransferase Increased (Gastrointestinal disorders) | 0 | 0 | 7
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 0 | 7
Blurred Vision (Eye disorders) | 0 | 0 | 7
Anorexia (Metabolism and nutrition disorders) | 12 | 0 | 0
Body Odor (General disorders) | 12 | 0 | 0
Breast Infection (Infections and infestations) | 12 | 0 | 0
Dehydration (General disorders) | 12 | 0 | 0
Erythema Multiforma (Skin and subcutaneous tissue disorders) | 12 | 0 | 0
Fever (General disorders) | 12 | 0 | 7
Febrile Neutropenia (Immune system disorders) | 12 | 0 | 0
Insomnia (General disorders) | 12 | 0 | 0
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 0 | 0
Pruitus (Skin and subcutaneous tissue disorders) | 12 | 0 | 0
Weight Loss (Metabolism and nutrition disorders) | 12 | 0 | 7
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes